## STATISTICAL ANALYSIS PLAN

**VERSION**: 1.4 **DATE**: 16-DEC-2020

#### **STUDY DRUG:**

Recombinant Crisantaspase Pseudomonas fluorescens (RC-P), JZP-458

#### PROTOCOL/STUDY NUMBER:

JZP458-201 Protocol original version (29 August 2019)
Amendment 01 (18 August 2020)
Amendment 02 (03 September 2020)

#### **STUDY TITLE:**

An Open-Label, Multicenter Study of RC-P in Patients with Acute Lymphoblastic Leukemia (ALL)/Lymphoblastic Lymphoma (LBL) Following Hypersensitivity to *E. coli*-derived *Asparaginases* 

## **SPONSOR (UNITED STATES REPRESENTATIVE):**

Jazz Pharmaceuticals
3170 Porter Dr, Palo Alto, CA 94304

This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

## **SIGNATURE PAGE**

This document has been prepared by:

Dir, Biostatistics Jazz Pharmaceuticals, Inc.

Dec-16-2020 | 10:56 AM PS

Date

This document has been reviewed and approved per the SOP by:

Dir, Biostatistics

Jazz Pharmaceuticals, Inc.

Dir, Clinical Pharmacology Jazz Pharmaceuticals, Inc.

Ex. Medical Director, Clinical Development Jazz Pharmaceuticals, Inc.

Dec-16-2020 | 10:56 AM PS7 Date Dec-16-2020 | 8:17 PM PST

Date

Dec-16-2020 | 11:45 AM PST

Date

## TABLE OF CONTENTS

| LIST OF | TABLES | 5 |
|---|---|---|
| LIST OF | FIGURES | 5 |
| LIST OF | APPENDICES | 5 |
| 1. | LIST OF ABBREVIATIONS | 6 |
| 2. | MODIFICATION HISTORY | 8 |
| 3. | INTRODUCTION | 9 |
| 4. | STUDY OBJECTIVES AND ENDPOINTS | 10 |
| 4.1. | Study Objectives | 10 |
| 4.1.1. | Primary Objectives | 10 |
| 4.1.2. | Secondary Objective | 10 |
| 4.1.3. | Exploratory Objectives | 10 |
| 4.2. | Study Endpoints | 11 |
| 4.2.1. | Primary Endpoints | 11 |
| 4.2.2. | Secondary Endpoints | 11 |
| 4.2.3. | Exploratory Endpoints | 11 |
| 5. | STUDY DESIGN | 13 |
| 5.1. | Summary of Study Design | 13 |
| 5.2. | Study Treatment | 16 |
| 5.3. | Power and Sample Size Considerations | 16 |
| 5.4. | Randomization and Blinding | 17 |
| 5.5. | Interim Analysis | 17 |
| 6. | ANALYSIS SETS | 18 |
| 7. | GENERAL ASPECTS FOR STATISTICAL ANALYSIS | 19 |
| 7.1. | General Methods | 19 |
| 7.2. | Study Day 1 and Baseline Value Definitions | 19 |
| 7.2.1. | Study Day 1 | 19 |
| 7.2.2. | Baseline Value | 19 |
| 7.2.3. | Study Day | 19 |
| 7.2.4. | Visit Windows | 19 |
| 7.2.5. | Missing and Partial Data | 19 |
| 7.3. | Hypotheses Testing, Level of Significance and Multiplicity Adjustment | 20 |

| 7.4. | Subgroups and Subgroup Analyses | 20 |
|---|---|---|
| 7.5. | Changes to Planned Analyses | 20 |
| 8. | STUDY POPULATION SUMMARIES | 21 |
| 8.1. | Enrollment | 21 |
| 8.2. | Subject Disposition | 21 |
| 8.3. | Demographic and Baseline Characteristics | 21 |
| 8.4. | Medical History | 22 |
| 8.5. | Prior and Concomitant Medications | 22 |
| 8.6. | Protocol Deviations | 22 |
| 9. | EFFICACY | 23 |
| 9.1. | Primary Efficacy Endpoint and Analysis | 23 |
| 9.1.1. | Primary Efficacy Endpoint | 23 |
| 9.1.2. | Analysis of the Primary Efficacy Endpoint | 23 |
| 9.1.3. | Sensitivity Analyses | 23 |
| 9.1.4. | Subgroup Analyses | 23 |
| 9.2. | Secondary Efficacy Endpoints and Analyses | 23 |
| 9.2.1. | Key Secondary Efficacy Endpoint | 23 |
| 9.2.2. | Other Secondary Efficacy Endpoints | 24 |
| 9.2.3. | Sensitivity analyses | 24 |
| 9.2.4. | Subgroup Analyses | 24 |
| 9.3. | Exploratory Efficacy Endpoints and Analyses | 24 |
| 9.3.1. | Proportion of patients with the Last 48-hour NSAA level $\geq$ 0.1 IU/mL during the first course of IV administration of RC-P | 25 |
| 9.3.2. | Proportion of patients with the Last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P | |
| 9.3.3. | Proportion of patients with the Last 48-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P | 25 |
| 9.3.4. | Proportion of patients with the Last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P | 25 |
| 10. | SAFETY | 27 |
| 10.1. | Exposure | 27 |
| 10.1.1. | Extent of Exposure | |
| 10.1.2. | Treatment Compliance | 27 |
| 10.2. | Adverse Events | 27 |

| Adverse Events of Special Interest | 29 |
|---|---|
| Laboratory Assessments | 29 |
| Vital Signs | 29 |
| Other Safety Endpoints | 29 |
| PHARMACOKINETIC/PHARMACODYNAMIC ANALYSES | 30 |
| IMMUNOGENICITY | 31 |
| COVID-19 | 32 |
| NCES | 32 |
| IX I. DATE IMPUTATION RULES | 33 |
| IX II. PTS USED TO SEARCH AES OF SPECIAL INTEREST | 35 |
| LIST OF TABLES | |
| List of Abbreviations | 6 |
| List of Abbreviations | 6 |
| (a) Part A IM RC-P Dose Cohorts; (b) Part B IV RC-P Dose Cohorts | 15 |
| LIST OF APPENDICES | |
| IX I. DATE IMPUTATION RULES | 33 |
| IX II. PTS USED TO SEARCH AES OF SPECIAL INTEREST | 35 |
| | List of Abbreviations List of Abbreviations List of Abbreviations List of Abbreviations List OF APPENDICES X I. DATE IMPUTATION RULES List OF APPENDICES X I. DATE IMPUTATION RULES LIST OF APPENDICES |

## 1. LIST OF ABBREVIATIONS

**Table 1:** List of Abbreviations

| Abbreviation | Term |
|--------------|---------------------------------------------------------------|
| ADA | Anti-drug antibody |
| AE | Adverse event |
| ALL | Acute lymphoblastic leukemia |
| BSA | Body surface area |
| CI | Confidence interval |
| COG | Children's Oncology Group |
| CSR | Clinical study report |
| CTCAE | Common terminology criteria for adverse events |
| CV | Coefficient of variation |
| E. coli | Escherichia coli |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| FDA | Food and Drug Administration |
| ICH | International Council for Harmonisation |
| IM | Intramuscular |
| IU | International unit(s) |
| LBL | Lymphoblastic lymphoma |
| IV | Intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NSAA | Nadir serum asparaginase activity |
| PD | Pharmacodynamics |
| PK | Pharmacokinetic |
| PT | Preferred term |
| RC-P | Recombinant crisantaspase produced in Pseudomonas fluorescens |
| SAA | Serum asparaginase activity |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDRC | Study data review committee |
| SOC | System organ class |

| SOP | Standard operating procedures |
|------|----------------------------------|
| TEAE | Treatment emergent adverse event |
| WHO | World Health Organization |

## 2. MODIFICATION HISTORY

Version History for SAP:

| Version | Date | Description |
|---|---|---|
| 1.0 | 18DEC2019 | Original |
| 1.1 | 07APR2020 | Clarification on the Efficacy/PK/PD |
| | | Analysis Sets and sample size at the |
| | | interim analysis in Section 5.3 |
| 1.2 | 08JUN2020 | Further clarification and language |
| | | update on the sample size at the interim |
| | | analysis in Section 5.3 |
| 1.3 | 24SEP2020 | <ul> <li>Update study design in Section 5 per protocol amendment 1 and 2.</li> <li>Clarification on the sample size at the primary analysis in Section 5.3.</li> <li>Addition of the sensitivity analyses to assess COVID-19 impact on the primary (Section 9.1.3) and key secondary (Section 9.2.3) efficacy endpoints.</li> </ul> |
| | | Addition of Section 13. COVID-19 |
| 1.4 | 16DEC2020 | • Added the term of pulmonary embolism to the list of preferred terms for the AE of special interest of thrombosis. |

#### 3. INTRODUCTION

This is an open-label, multicenter, dose confirmation, and pharmacokinetic (PK) study of Recombinant Crisantaspase Produced in *Pseudomonas fluorescens* (RC-P) in patients (of any age) with acute lymphoblastic leukemia (ALL)/lymphoblastic lymphoma (LBL) who are hypersensitive to *E. coli*-derived asparaginases (allergic reaction or silent inactivation).

This study has *i*) one interim analysis which is planned after the 51<sup>st</sup> patient completes Course 1 at the final intramuscular (IM) RC-P dose in Part A (Cohorts 1 and 2), *ii*) one primary analysis which is planned after the 98<sup>th</sup> patient completes Course 1 at the final IM RC-P dose in Part A (Cohorts 1 and 2), and *iii*) the final analysis which is planned when the overall study (Part A and Part B) is complete and all enrolled patients have completed all of their planned courses of RC-P, including end of study procedures, or have discontinued the study early.

The purpose of this statistical analysis plan (SAP) is to describe in detail the statistical methodology and planned analyses to be conducted for the interim, primary and final analysis of Protocol JZP458-201 for inclusion in the Clinical Study Report (CSR). The current version is based on Protocol amendment 02 dated 03 September 2020. Any additional analyses or deviation from the analyses outlined in this plan will be documented with rationale in the final clinical study report (CSR).

#### 4. STUDY OBJECTIVES AND ENDPOINTS

## 4.1. Study Objectives

#### 4.1.1. Primary Objectives

The primary objectives of the study are as follows:

- To determine the efficacy of intramuscular (IM) RC-P administration as measured by the response in Cohort 1 and Cohort 2, defined as the last 72-hour nadir serum asparaginase activity (NSAA) level ≥ 0.1 IU/mL during the first course
- To assess the safety and tolerability of IM RC-P in patients with ALL/LBL who are hypersensitive to *E. coli*-derived asparaginases

### 4.1.2. Secondary Objective

#### 4.1.2.1. Key Secondary Objective

The key secondary objective of the study is to determine the efficacy of IM RC-P administration as measured by the response in Cohort 1 and Cohort 2, defined as the last 48-hour NSAA level  $\geq 0.1 \text{ IU/mL}$  during the first course.

#### 4.1.2.2. Secondary Objectives

Other secondary objectives of the study are as follows:

- To determine the efficacy of IM RC-P administration as measured by the response in Cohort 1 and Cohort 2, defined as the last 48-hour and the last 72-hour NSAA levels ≥ 0.4 IU/mL during the first course
- To characterize the pharmacokinetics (PK) of IM RC-P using a population PK approach, and to explore exposure-response correlations
- To assess the immunogenicity of IM RC-P following repeat administration of RC-P

#### 4.1.3. Exploratory Objectives

The exploratory objectives of this study are as follows:

- To determine the efficacy of intravenous (IV) RC-P administration as measured by the response, defined as the last 48-hour NSAA ≥ 0.1 IU/mL and the last 72-hour NSAA ≥ 0.1 IU/mL during the first course
- To determine the efficacy of IV RC-P administration measured by the response, defined as the last 48-hour NSAA ≥ 0.4 IU/mL and the last 72-hour NSAA ≥ 0.4 IU/mL during the first course
- To assess the safety and tolerability of IV RC-P in patients with ALL/LBL who are hypersensitive to *E. coli*-derived asparaginases
- To characterize the PK of IV RC-P using a population PK approach
- To assess the immunogenicity of IV RC-P following repeat administration of RC-P

## 4.2. Study Endpoints

### 4.2.1. Primary Endpoints

- The primary efficacy endpoint of the study is the response rate, defined as the proportion of patients with the last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IM RC-P. Depending on the RC-P start day for a patient, this could be predose 4 if the first course of RC-P started on a Monday; predose 6 if the first course of RC-P started on a Wednesday; or predose 5 if the first course of RC-P started on a Friday.
- The primary safety endpoint of the study is the safety and tolerability of IM RC-P in patients with ALL/LBL who are hypersensitive to *E. coli*-derived asparaginases. This swill be determined by the occurrence of treatment-emergent adverse events.

#### 4.2.2. Secondary Endpoints

#### 4.2.2.1. Key Secondary Endpoint

• Proportion of patients with the last 48-hour NSAA level ≥ 0.1 IU/mL during the first course of IM administration of RC-P

#### 4.2.2.2. Other Secondary Endpoints

Secondary endpoints for patients in Part A:

- Proportion of patients with the last 48-hour NSAA level ≥ 0.4 IU/mL during the first course of IM administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IM administration of RC-P
- Characterization of the PK of IM RC-P based on SAA using a population PK approach and exposure-response correlations
- Incidence of anti-drug antibody (ADA) formation against RC-P

#### 4.2.3. Exploratory Endpoints

Exploratory endpoints for patients in Part B:

- Proportion of patients with the last 48-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 48-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P
- Incidence of treatment emergent adverse events
- Characterization of the PK of IV RC-P based on SAA using a population PK approach

• Incidence of ADA formation against RC-P

## 5. STUDY DESIGN

## 5.1. Summary of Study Design

This study is designed to assess the tolerability and efficacy of RC-P (only in patients with ALL/LBL who develop hypersensitivity to an *E. coli*-derived asparaginase), as measured by asparaginase activity. In this patient population, 6 doses of RC-P should be substituted for each dose of a long-acting *E. coli*-derived asparaginase. Two consecutive weeks' treatment of RC-P is defined as one course. Additional courses of RC-P will be administered based on each patient's original treatment plan for as long as the patient derives clinical benefit.

This study will consist of two parts: **Part A** to determine the dose of RC-P for IM administration and to confirm safety and efficacy; and **Part B** to define the optimal dose and schedule of IV RC-P. Part A and Part B may be investigated in parallel.

Efficacy and safety data will be assessed by a Study Data Review Committee (SDRC) at frequent intervals as described below. The SDRC will make recommendations and have oversight of the study as described in the protocol and the SDRC Charter. The SDRC will review results throughout the study as follows: for Part A at n = 6 and 13 (for each Cohort 1 subcohort), at n = 19, 32, and 51 (Cohort 1 plus Cohort 2 at the final IM RC-P dose with n=51 as the interim analysis); and Part B at n = 6 at a minimum.

#### **IM RC-P Dose Confirmation (Part A):**

Part A (IM RC-P) of the study will have 2 IM cohorts:

- Cohort 1 (includes multiple subcohorts), an RC-P repeat dose/confirmatory cohort with the initial RC-P dose of 25 mg/m<sup>2</sup> based on data from the Phase 1 healthy subject study; a final IM RC-P dose level will be selected, and
- Cohort 2, an expansion cohort to confirm the efficacy and safety of the final IM RC-P dose level and schedule; a maximum target of 20% of the patients enrolled in Cohort 2 may enter the study based on a Grade 2 allergic reaction (Inclusion Criterion #3).

**Part A Cohort 1 (IM Dose Confirmation):** Patients in this cohort will be administered 6 doses of IM RC-P (Course 1), to evaluate the safety/tolerability and efficacy of repeated doses of IM RC-P. Cohort 1 patients will have 6 IM RC-P doses administered on a Monday, Wednesday, Friday (MWF) schedule over 2 weeks with the initial dose starting either on a Monday or Wednesday or Friday (depending on the patient's planned chemotherapy schedule). The starting dose for RC-P Dose Cohort 1a will be 25 mg/m<sup>2</sup>. Additional subcohorts (eg, Cohort 1b, Cohort 1c...Cohort 1x) may be enrolled to determine the optimal dose for Cohort 2.

A target of 13 evaluable patients will be enrolled in each Cohort 1 subcohort. Evaluable patients for Cohort 1 are defined as patients who have received at least 3 doses of IM RC-P and have a 72-hour NSAA level (obtained within  $\pm$  2-hour window) during the second half of Course 1. For patients who are treated but are not evaluable, additional patients may be enrolled. Patients who discontinue RC-P will be evaluated for safety.

The SDRC will review the data when 6 evaluable patients in each subcohort complete Course 1. If 6 of the 6 evaluable patients in that subcohort have a 72-hour NSAA level  $\geq$  0.1 IU/mL and the safety/tolerability issues are acceptable based on a review by the SDRC, then the SDRC will also review the data when 13 evaluable patients in each subcohort complete Course 1. If 13 of the 13 (100%) evaluable patients in that subcohort have 72-hour NSAA levels  $\geq$  0.1 IU/mL and the safety/tolerability issues are acceptable based on a review by the SDRC, no additional patients will be enrolled in Cohort 1. Patients will be enrolled at this IM RC-P dose level in Part A Cohort 2 of this study.

If 1 or more of the 13 evaluable patients in the subcohort has a 72-hour NSAA level < 0.1 IU/mL, or if any safety/tolerability issues are not acceptable based on a review by the SDRC, then the PK and safety data will be analyzed to determine whether a new subcohort (with a lower dose, higher dose, or different doses on different days) is needed. Based on all of the data, the SDRC may recommend that a different dose be given on Fridays than on Mondays and Wednesdays. Any additional dose level(s) studied for RC-P will not exceed a 50% increase from the previous dose level.

**Part A Cohort 2 (IM Expansion):** Approximately 85 patients are expected to be enrolled in this cohort and each patient is planned to receive at least 6 doses (1 course) of IM RC-P at the final IM RC-P dose level selected from Part A Cohort 1.

The SDRC will review the data on NSAA levels at frequent intervals for Cohort 2; these reviews will occur when totals of 19, 32, and 51 patients (Cohort 1 plus Cohort 2 at the final IM RC-P dose with n=51 as the interim analysis) complete Course 1. In addition, the SDRC will review the data to assess the safety of the selected dose level when 32 and 51 patients complete Course 1. Enrollment for this cohort may be stopped if the incidence of allergic reactions (including hypersensitivity and anaphylaxis) related to RC-P exceeds 25%, or the incidence of pancreatitis exceeds 10% or thrombosis exceeds 10%.

#### **IV RC-P Dose Confirmation (Part B):**

Part B (IV RC-P) may begin in parallel with Part A; study center participation will be at the discretion of the Sponsor. Part B of this study will be conducted to define the optimal dose of the IV administration of RC-P for further study in ALL/LBL patients as a repeated dose. Part B patients will have 6 IV RC-P doses administered on a MWF schedule over 2 weeks with the initial dose starting either on a Monday or Wednesday or Friday (depending on the patient's planned chemotherapy schedule).

Part B (IV RC-P) of the study will have at least 1 IV subcohort at a starting dose of 37.5 mg/m<sup>2</sup>:

• Cohort 1 (may include multiple subcohorts), IV RC-P Dose Confirmation

**Part B Cohort 1 (IV Dose Confirmation):** RC-P to study IV administration in Part B Cohort 1 will be provided as 6 doses for each patient.

A target of at least 6 evaluable patients will be enrolled in Cohort 1a; more patients may be enrolled as described below. Evaluable patients for Cohort 1 are defined as patients who have received at least 3 doses of IV RC-P and have a 72-hour NSAA level (obtained within the  $\pm$  2-

hour window) during the second half of Course 1. For patients who are treated but are not evaluable, additional patients may be enrolled.

If 6 of the 6 evaluable patients in Cohort 1a have a 72-hour NSAA level  $\geq 0.1$  IU/mL and the safety/tolerability issues are acceptable based on a review by the SDRC, the dose may be confirmed as a dose for further evaluation. If the dose is not confirmed, additional subcohorts may be investigated. The dose chosen for further evaluation may be used in a Part B IV expansion cohort of this study using a similar design as used in Part A Cohort 2, if the Sponsor determines that an IV Expansion Cohort 2 is to be done in this study (Figure 1b).

Figure 1: (a) Part A IM RC-P Dose Cohorts; (b) Part B IV RC-P Dose Cohorts



### **5.2.** Study Treatment

Dosages (mg/m²) will be administered based on the patient's body surface area (BSA), and calculated using the patient's height and weight taken prior to the start of each course. Patients will receive doses of either RC-P via the IM or IV route depending on whether they are enrolled in Part A (IM) or Part B (IV) of the study. All other chemotherapy will continue according to the therapeutic regimen as defined in the patient's original treatment protocol for the patient's ALL/LBL.

In Part A of the study, RC-P will be administered via the IM route. For IM RC-P Dose Cohort 1, the starting dose of RC-P will be 25 mg/m<sup>2</sup> with 6 IM RC-P doses.

In Part B of the study, RC-P will be administered via the IV route. For IV RC-P Dose Cohort 1, the starting dose of RC-P is planned to be  $37.5 \text{ mg/m}^2$  with 6 IV RC-P doses.

## **5.3.** Power and Sample Size Considerations

For Part A of the study, 98 patients administered the final IM dose level are planned.

For the final IM RC-P dose level, 13 evaluable patients are planned in Part A Cohort 1 (IM RC-P Dose Confirmation), and approximately 85 patients are planned in Cohort 2 (IM Expansion) to obtain 98 patients in total at the final dose in Part A for the primary efficacy analysis of the IM administration route.

The sample size of 13 evaluable patients in Part A Cohort 1 provides at least 80% posterior probability of the true response rate  $\geq 96\%$  given 100% response rate in Cohort 1 and non-informative neutral beta prior with  $\alpha = \beta = 1/3$ .

Since the primary efficacy endpoint is considered to be met if the lower bound of the 95% Wald confidence interval (CI) of the response rate exceeds 90%, the final sample size is planned as 98 patients which provides 83% probability that the lower bound of the 95% Wald CI exceeds 90%, assuming a true response rate of 96% for the primary efficacy endpoint and a 5% drop out rate. Furthermore, with a sample size of 98 patients, the probability of observing at least one adverse events (AE) related to asparaginase with an incidence as low as 3% is 95%.

For the primary efficacy assessment at the primary analysis, a minimum of 93 patients in the Efficacy Analysis Set are required. This means at least 93 patients received at least one dose of the final IM RC-P dose level, and had at least one 72-hour NSAA assessment collected within the protocol-defined sample collection window (± 2 hours) in Course 1. If fewer than 93 out of 98 patients have the necessary data, additional patients will be enrolled to ensure 93 patients for analysis.

One interim analysis with 51 patients is planned. At the interim analysis, a sample size of 51 patients provides 70% probability that the lower bound of the 95% CI exceeds 90% under the assumption of a 96% true response rate and a 5% drop out rate. The probability of observing at least one AE related to asparaginase with an incidence as low as 3% is 79% with 51 patients.

Similar to the primary analysis, a minimum of 48 patients in the Efficacy Analysis Set for the primary efficacy assessment are necessary for the interim analysis. If fewer than 48 out of 51 patients have the necessary data, additional patients will be enrolled to ensure 48 patients for analysis.

For Part B, a target of at least 6 evaluable patients will be administered the first IV dose level. This sample size is not based on formal power calculation but provides an initial assessment of the IV RC-P dosing.

## 5.4. Randomization and Blinding

This is an open-label study; there will be no blinding. Participants to the study will not be randomized.

## 5.5. Interim Analysis

This study has one interim analysis planned after the 51<sup>st</sup> patient completes Course 1 with the final IM RC-P dose level (Cohort 1 and Cohort 2 patients). If the primary endpoint is met at the interim analysis, the enrollment to this cohort will be stopped early for efficacy. If the incidence of allergic reactions (including hypersensitivity and anaphylaxis) related to RC-P exceeds 25%, or the incidence of pancreatitis exceeds 10% or thrombosis exceeds 10% at this interim analysis, enrollment into this Expansion Cohort may be stopped for safety.

Page 17 of 45

## 6. ANALYSIS SETS

For purposes of analysis, the following populations are defined.

| Analysis Set | Description |
|---|---|
| Enrolled Analysis Set | The Enrolled Analysis Set includes patients who signed the informed consent and meet inclusion/exclusion criteria per investigator. |
| Efficacy Analysis Set | The Efficacy Analysis Set includes patients who received at least one dose of RC-P and had at least one 48- or 72-hour NSAA assessment collected within the protocol defined sample collection window (± 2 hours) in Course 1. This will be the primary analysis set for the primary efficacy endpoint and all other efficacy endpoints. |
| Safety Analysis Set | The Safety Analysis Set will include patients who received at least one dose of RC-P. This will be the primary analysis set for the primary safety endpoint and all other safety endpoints. |
| PK Analysis Set | The PK Analysis Set will include patients who received at least one dose of RC-P and have at least one post-dose evaluable SAA or PK concentration value. This will be used for all descriptive PK summaries. |
| PD Analysis Set | The Pharmacodynamics (PD) Analysis Set will include patients who received at least one dose of RC-P and have at least one post-dose evaluable L-asparagine or L-glutamine value. This will be used for all descriptive PD summaries. |

#### 7. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

The statistical principles applied in the design and planned analyses of this study are consistent with International Conference for Harmonisation (ICH) E9 guidelines (ICH 1998).

#### 7.1. General Methods

Unless otherwise specified, continuous data will be summarized using descriptive statistics comprising of the number of patients with data to be summarized (n), mean, standard deviation (SD), median, minimum (min) and maximum (max), by time, dose level of RC-P, and route of administration (IM or IV) as appropriate. Categorical variables will be presented using counts and percentages.

Unless otherwise specified, analyses and summary outputs will be generated using SAS® version 9.4 (or higher).

## 7.2. Study Day 1 and Baseline Value Definitions

#### **7.2.1.** Study Day 1

Study Day 1 is defined as the date of the first dose of RC-P.

#### 7.2.2. Baseline Value

A baseline value is defined as the latest non-missing value obtained prior to or at the start date and/or time of the first dose of RC-P.

#### **7.2.3. Study Day**

Study Day is calculated relative to Study Day 1 as follows:

- If the date of the event is on or after Study Day 1, Study Day = (date of event - Study Day 1) +1.
- If the date of the event is prior to Study Day 1,
   Study Day = (date of event Study Day 1).

#### 7.2.4. Visit Windows

Not applicable.

#### 7.2.5. Missing and Partial Data

Any missing AE information such as severity and relationship will be handled as described in Section 10.2 and Appendix I.

Missing PK levels will be handled as described in Section 11.

# 7.3. Hypotheses Testing, Level of Significance and Multiplicity Adjustment

No formal statistical testing is planned for this study and thus no multiplicity adjustment is applicable.

## 7.4. Subgroups and Subgroup Analyses

Exploratory analyses of the primary efficacy, secondary efficacy, and safety endpoints may be conducted for the following subgroups of interest:

- Pediatric (<18) vs adult ( $\ge 18$ )
- Patients with prior allergic reaction to an *E. coli*-derived asparaginase vs silent inactivation
- Patients with Grade 2 allergic reaction vs Grade 3 allergic reactions

## 7.5. Changes to Planned Analyses

Sensitivity analyses were added to assess COVID-19 impact on the primary (Section 9.1.3) and key secondary (Section 9.2.3) efficacy endpoint. Additional subgroup analyses for the primary (Section 9.1.4) and secondary (Section 9.2.4) efficacy endpoints which are not specified in the protocol may be performed.

Summary of protocol deviations due to COVID-19 was newly added in Section 13.

#### 8. STUDY POPULATION SUMMARIES

#### 8.1. Enrollment

Listings of inclusion/exclusion criteria for enrollment will be provided.

## 8.2. Subject Disposition

The summary of patient disposition will include the number of patients screened, screen failure patients who were not enrolled with summary of reasons, patients in the Enrolled Analysis Set, and patients in the following categories:

## **Study Drug Completion**

- Received at least one dose of study drug treatment
- Ongoing study drug treatment
- Completed study drug treatment
- Discontinued study drug treatment with summary of reasons for discontinuing study drug treatment

#### **Study Completion**

- Ongoing study
- Completed study
- Discontinued study with summary of reasons for discontinuing study

This summary will be provided by dose level of RC-P and route of administration (IM or IV).

A separate summary of the study analysis sets will be provided to include the number of patients in the Enrolled Analysis Set, patients in the Efficacy Analysis Set, patients in the Safety Analysis set, patients in the PK Analysis Set, and patients in PD Analysis Set.

A listing of patient disposition with study analysis set, study drug completion and study completion status will be provided.

## 8.3. Demographic and Baseline Characteristics

Patient demographics (e.g. gender, race, ethnicity, and age at enrollment) and baseline characteristics (e.g. weight, height, body mass index [BMI], and BSA) will be summarized by dose level of RC-P and route of administration (IM or IV) for the Efficacy, Safety, and PK Analysis Sets. A listing of demographic and baseline characteristics will be provided for Safety Analysis Set.

In addition, the following baseline characteristics and medical history will be summarized:

- Primary disease (ALL vs LBL)
- Time since primary disease diagnosis to Study Day 1
- Prior asparaginase treatment
- Time since last asparaginase received to Study Day 1

• Prior Grade 2 vs Grade 3 allergic reaction to an E. coli-derived asparaginase vs silent inactivation

No formal statistical comparisons will be performed.

## 8.4. Medical History

Medical history will be coded using the MedDRA 22.1 and listed by dose level of RC-P, route of administration (IM or IV), system organ class (SOC), and preferred term (PT) for Safety Analysis Set. For data presentation, SOC will be ordered alphabetically, with PT sorted by decreasing frequency in the final dose of IM.

#### 8.5. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary and will be summarized separately by dose level of RC-P and route of administration (IM or IV) for the Safety Analysis Set.

Prior medications are defined as those medications taken prior to Study Day 1. Concomitant medications are defined as medications taken at any time on or after Study Day 1. If any medications were taken prior to Study Day 1 and continued to or after Study Day 1, it will be counted as both prior and concomitant medications. Like AEs, prior and concomitant definitions for medications will be derived after taking into consideration any partial or completely missing start and end dates (See Appendix I).

Listings of prior medications and concomitant medications will be provided separately.

#### **8.6.** Protocol Deviations

Major protocol deviations will be summarized by dose level of RC-P and route of administration (IM or IV) using the Safety Analysis Set. All protocol deviations will be listed.

#### 9. EFFICACY

## 9.1. Primary Efficacy Endpoint and Analysis

#### 9.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint of the study is the response rate, defined as the proportion of patients with the last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IM administration of RC-P. Patients in both Part A Cohort 1 and Cohort 2 at the final IM RC-P dose level will be included. Depending on the RC-P start day for a patient, this could be predose 4 if the first course of RC-P started on a Monday; predose 6 if the first course of RC-P started on a Wednesday; or predose 5 if the first course of RC-P started on a Friday.

#### 9.1.2. Analysis of the Primary Efficacy Endpoint

The primary efficacy endpoint will be estimated using the Efficacy Analysis Set for patients administered the final IM RC-P dose level with at least one 72-hour NSAA assessment collected within the protocol defined sample collection window (± 2 hours) in Course 1 of Part A. The last observed 72-hour NSAA assessment collected within the protocol defined sample collection window (± 2 hours) in Course 1 will be used in the calculation of the primary efficacy endpoint. Missing data will not be imputed. The response rate, along with the 95% Wald CI will be provided. The primary efficacy endpoint will be met if the lower bound of the 95% CI of the response rate exceeds 90%.

#### 9.1.3. Sensitivity Analyses

A sensitivity analysis will be performed to assess COVID-19 impact on the primary efficacy endpoint. Patients in the Efficacy Analysis Set who missed any PK sample collections in Course 1 due to COVID-19 will be excluded from the analysis. The response rate for this subset along with the 95% Wald CI will be provided.

#### 9.1.4. Subgroup Analyses

The primary efficacy endpoint will be analyzed for the patient subgroups specified in Section 7.4.

## 9.2. Secondary Efficacy Endpoints and Analyses

#### 9.2.1. Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint of the study is the response rate, defined as the proportion of patients with the last 48-hour NSAA level  $\geq$  0.1 IU/mL during the first course of IM administration of RC-P.

The key secondary efficacy endpoint will be analyzed using the Efficacy Analysis Set for patients administered the final IM RC-P dose level with at least one 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part A. The last observed 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of the key secondary efficacy endpoint. Missing data will not be imputed. The response rate, along with the 95% Wald CI will

be provided. The key secondary efficacy endpoint will be met if the lower bound of the 95% CI of the response rate exceeds 90%.

#### 9.2.2. Other Secondary Efficacy Endpoints

Other secondary efficacy endpoints in Part A include the following:

- Proportion of patients with the last 48-hour NSAA level ≥ 0.4 IU/mL during the first course of IM administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IM administration of RC-P

# 9.2.2.1. Proportion of Patients with the Last 48-hour NSAA Level ≥ 0.4 IU/mL during the First Course of IM Administration of RC-P

The proportion of patients with the last 48-hour NSAA level  $\geq 0.4$  IU/mL during the first course of IM administration of RC-P will be analyzed using the Efficacy Analysis Set for patients administered the final IM RC-P dose level with at least one 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part A. The last observed 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% Wald CI will be provided.

# 9.2.2.2. Proportion of Patients with the Last 72-hour NSAA Level ≥ 0.4 IU/mL during the First Course of IM Administration of RC-P

The proportion of patients with the last 72-hour NSAA level  $\geq 0.4$  IU/mL during the first course of IM administration of RC-P will be analyzed using the Efficacy Analysis Set for patients administered the final IM RC-P dose level with at least one 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part A. The last observed 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% Wald CI will be provided.

#### 9.2.3. Sensitivity analyses

A sensitivity analysis will be performed to assess COVID-19 impact on the key secondary efficacy endpoint. Patients in the Efficacy Analysis Set who missed any PK sample collections in Course 1 due to COVID-19 will be excluded from the analysis. The response rate for this subset along with the 95% Wald CI will be provided.

#### 9.2.4. Subgroup Analyses

The key and other secondary efficacy endpoints will be analyzed for the patient subgroups specified in Section 7.4.

## 9.3. Exploratory Efficacy Endpoints and Analyses

Exploratory efficacy endpoints include the following from Part B of the study:

- Proportion of patients with the last 48-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 48-hour NSAA levels ≥ 0.4 IU/mL during the first course of IV administration of RC-P
- Proportion of patients with the last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P

# 9.3.1. Proportion of patients with the Last 48-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P

The proportion of patients with the last 48-hour NSAA level  $\geq 0.1$  IU/mL during the first course of IV administration of RC-P will be analyzed using the Efficacy Analysis Set for patients administered the final IV RC-P dose level with at least one 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part B. The last observed 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% CI will be provided.

# 9.3.2. Proportion of patients with the Last 72-hour NSAA level ≥ 0.1 IU/mL during the first course of IV administration of RC-P

The proportion of patients with the last 72-hour NSAA level  $\geq 0.1$  IU/mL during the first course of IV administration of RC-P will be analyzed using the Efficacy Analysis Set for patients administered the final IV RC-P dose level with at least one 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part B. The last observed 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% CI will be provided.

# 9.3.3. Proportion of patients with the Last 48-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P

The proportion of patients with the last 48-hour NSAA level  $\geq 0.4$  IU/mL during the first course of IV administration of RC-P will be analyzed using the Efficacy Analysis Set for patients administered the final IV RC-P dose level with at least one 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part B. The last observed 48-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% CI will be provided.

# 9.3.4. Proportion of patients with the Last 72-hour NSAA level ≥ 0.4 IU/mL during the first course of IV administration of RC-P

The proportion of patients with the last 72-hour NSAA level  $\geq 0.4$  IU/mL during the first course of IV administration of RC-P will be analyzed using the Efficacy Analysis Set for patients

administered the final IV RC-P dose level with at least one 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 of Part B. The last observed 72-hour NSAA assessment collected within the protocol defined sample collection window ( $\pm$  2 hours) in Course 1 will be used in the calculation of this endpoint. Missing data will not be imputed. The response rate, along with the 95% CI will be provided.

#### 10. SAFETY

Safety analyses will be summarized by dose level of RC-P, and route of administration (IM or IV) using the Safety Analysis Set. No formal statistical testing will be performed for the safety analyses.

### 10.1. Exposure

#### 10.1.1. Extent of Exposure

The summary of *i*) planned and actual RC-P administration status by course, and *ii*) the descriptive summary of planned and actual number of courses of RC-P will be provided. Study drug administration details such as the course number, actual dose, start and end day/time of the study drug administration will be listed separately.

#### **10.1.2.** Treatment Compliance

Not applicable for this study since RC-P administration will vary depending on the number of doses of a long-acting *E. coli*-derived asparaginase remaining on an individual patient's original treatment protocol.

#### 10.2. Adverse Events

AEs recorded in the case report form will be coded to system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA 22.1). The investigator will assess the relatedness of each AE to study drug. The severity of AEs will be recorded using the Common Terminology Criteria for Adverse Events (CTCAE 5.0).

At a minimum, the investigator must record all AEs that occur from the time written informed consent is obtained until screen failure if applicable, or 30 days after the patient's last dose of the last course of RC-P, regardless of their relationship to study drug. Any serious AE (SAE) assessed as related to study drug by the investigator that occurs more than 30 days after the patient's last dose of the last course of RC-P should be reported regardless of time after study termination.

A treatment-emergent adverse event (TEAE) is defined as any event with onset date on or after Study Day 1 through the end of the study or any ongoing event that worsens in severity after Study Day 1 through the end of the study. Only TEAEs with the onset date through the end of the AE reporting period will be included in summary tables unless otherwise specified. For the purpose of calculating treatment emergence, incomplete onset dates will be imputed as detailed in Appendix I.

AEs are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe or medically significant but not immediately life-threatening), Grade 4 (life-threatening consequences), or Grade 5 (Death related to AE). The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings, and will be considered the least severe for the purposes of sorting for data presentation.

Treatment-related AEs are those for which the investigator answers "Yes" to the question "Was this adverse event related to study treatment?" in the eCRF. Events for which the investigator did not record relationship to study treatment will be considered related to study treatment for summary purpose. Data listings will show treatment-relationship as missing. AEs for which "Yes"

is marked for question "Was this adverse event related to study procedure?" in eCRF will be identified and included in AE listing.

SAEs are those for which the investigator answers "Yes" to the question "Was the adverse event serious?" in the eCRF. The clinical database will be reconciled with the SAE database before database finalization.

For all AE summaries, if a patient has more than 1 AE within a PT, the patient is counted only once at the maximum severity and with the closest relationship to study drug. If a patient has more than 1 AE within a SOC, the patient is similarly counted once when reporting results for that SOC.

A brief summary of TEAEs (i.e., the number and percentage of patients) will be presented by dose level of RC-P, and route of administration (IM or IV) for the following: (1) any TEAE, (2) any serious TEAE, (3) any treatment-related TEAE, (4) any serious treatment-related TEAE, (5) any Grade 3 or 4 TEAE, (6) any treatment-related Grade 3 or 4 TEAE, (7) any TEAE leading to study drug discontinuation, (8) any treatment-related TEAE leading to study drug discontinuation, (9) any TEAE leading to death, and (10) any treatment-related TEAE leading to death.

A general summary of TEAEs by SOC and PT will be provided with the number and percent of patients who experienced the following types of events by dose level of RC-P, and route of administration (IM or IV). For data presentation, SOC will be ordered alphabetically, with PT sorted by decreasing frequency in the final dose of IM:

- Patients with any TEAE
- Patients with any serious TEAE
- Patients with any treatment-related TEAE
- Patients with any serious treatment-related TEAE
- Patients with any Grade 3 or 4 TEAE
- Patients with any treatment-related Grade 3 or 4 TEAE
- Patients with any TEAE leading to study drug discontinuation
- Patients with any treatment-related TEAE leading to study drug discontinuation
- Patients with any TEAE leading to death
- Patients with any treatment-related TEAE leading to death

Data listings will be provided for the following including patient number, dose level of RC-P, route of administration (IM or IV), SOC, PT, date of onset/stop, severity, seriousness, treatment-relationship, action taken:

- All AEs
- Serious AEs
- Treatment-related AEs
- Serious treatment-related AEs
- Grade 3 and 4 AEs

- AEs leading to study drug discontinuation
- Death report

### 10.2.1. Adverse Events of Special Interest

AEs of special interest - allergic reactions (including hypersensitivity and anaphylaxis), pancreatitis, and thrombosis - will be summarized by dose level of RC-P, route of administration (IM or IV), and patients subgroups specified in Section 7.4. The list of PTs used to search each AEs of special interest, reviewed by Jazz Drug Safety & Pharmacovigilance, is provided in Appendix II.

## 10.3. Laboratory Assessments

Baseline value, post-baseline value, and changes from baseline value for all hematology, coagulation, and chemistry parameters will be summarized by dose level of RC-P and route of administration (IM or IV) using descriptive statistics.

## 10.4. Vital Signs

Baseline value, post-baseline value, and changes from baseline value for all vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate) and body temperature will be summarized by dose level of RC-P and route of administration (IM or IV) using descriptive statistics.

## 10.5. Other Safety Endpoints

A data listing will be provided for patients experiencing pregnancy during the study.

#### 11. PHARMACOKINETIC/PHARMACODYNAMIC ANALYSES

The summary and listings of RC-P PK (SAA and serum asparaginase concentration levels) and PD (asparagine and glutamine concentrations) measurements will be provided. Descriptive statistics including number of patients, mean, SD, median, min, max, coefficient of variation (CV), geometric mean, and geometric standard deviation will be used to summarize PK and PD data by time, dose level, Course, and route of administration (IM or IV), as appropriate. Proportion of patients with NSAA > 0.1 and > 0.4 IU/mL by time will also be summarized for SAA data.

Individual and/or summary figures of SAA-time or enzyme concentration-time profiles in serum may be provided. Individual and/or summary figures of SAA versus PD profiles may also be provided.

Statistical summaries and displays will be based on scheduled sampling times unless significant deviations occur (outside of the specified time windows in Appendix 2 in protocol). Differences between scheduled and actual sampling times will be listed for all patients.

RC-P SAA data will be used in a population PK analysis. A population PK model will be used to characterize the RC-P PK profiles in patients with ALL/LBL following hypersensitivity to *E. coli*derived asparaginases, and to explore exposure-response correlations. Results from the population PK analysis will be reported separately from the CSR, in a standalone document.

#### 12. IMMUNOGENICITY

The summary of immunogenicity results will be provided by dose level, Course, and route of administration (IM or IV) as appropriate. Immunogenicity results will be also listed as positive or negative for the presence of ADA for each patient by dose level, Course, and route of administration (IM or IV), as appropriate. In addition, for all ADA positive samples, titer values will be provided as a quantification measurement of antibodies.

For those with positive ADA results, individual profile may be provided to present ADA and hypersensitivity onset time along with each course start time. Boxplots of serum asparaginase activity levels by ADA status may also be provided.

#### 13. **COVID-19**

Data identifying missed visits, missed assessments, study drug discontinuation, and/or study participation termination due to COVID-19 will be captured either in EDC (study drug discontinuation and study participation termination) or protocol deviation log (missed visits and missed assessments). The collected data will specify if the study disruption was due to acquiring COVID-19 or due to other COVID-19 restrictions.

A summary of major protocol deviations due to COVID-19 will be provided. A listing of all disruptions due to COVID-19 will be provided (i.e. missed visits, missed assessments, study drug discontinuation, and study participation termination).

#### REFERENCES

Not applicable.

#### APPENDIX I. DATE IMPUTATION RULES

### Incomplete Adverse Event Onset Date

If *year* is missing (or completely missing): set to the date of first dose.

If (year is present and month and day are missing) or (year and day are present and month is missing):

If *year* = year of first dose: set the date to the first dose date.

If year < year of first dose: set month and day to December 31st.

If year > year of first dose: set month and day to January 1<sup>st</sup>.

If *month* and *year* are present and *day* is missing:

If *year* = year of first dose, and:

If *month* = month of first dose: set *day* to day of first dose.

If *month* < month of first dose: set *day* to last day of *month*.

If month > month of first dose: set day to  $1^{st}$  day of month.

If *year* < year of first dose: set *day* to last day of month.

If year > year of first dose: set day to 1<sup>st</sup> day of month.

For all other cases: set to date of first dose.

#### Incomplete Concomitant Medication Start Date

If *year* is missing (or completely missing): do not impute.

If (year is present and month and day are missing) or (year and day are present and month is missing):

Set *month* and day to January 1<sup>st</sup>.

If *year* and *month* are present and *day* is missing:

Set day to 1st day of month.

### <u>Incomplete Concomitant Medication End Date</u>

Do not impute if Ongoing Flag is checked.

If *year* is missing (or completely missing): do not impute.

If (year is present and month and day are missing) or (year and day are present and month is missing):

Set *month* and day to December 31<sup>st</sup>.

If *year* and *month* are present and *day* is missing:

Set *day* to last day of the month.

#### Incomplete Subsequent Anti-Leukemic/Cancer Therapy Start Date

Assumption: Anti-Cancer therapies reported on the Subsequent Anti-Leukemic/Cancer Therapy eCRF.

If *year* is missing (or completely missing): set to date of last dose of study treatment + 1 If (*year* is present and *month* and *day* are missing) or (*year* and *day* are present and *month* is missing):

If year > year of the last dose: Set *month* and day to January 1<sup>st</sup>.

If year = year of the last dose: Set month and day to date of last dose of study treatment + 1

If *year* and *month* are present and *day* is missing:

Set *day* to 1<sup>st</sup> day of month if the resulting imputed date is greater than date of last dose. Otherwise set the imputed date to date of last dose + 1

NOTE:If progressive disease/Relapse date is available and after date of last dose, replace last dose of study drug with progressive disease/Relapse date for imputation algorithm given in this section.

#### APPENDIX II. PTS USED TO SEARCH AES OF SPECIAL INTEREST

## List of PTs under the narrow SMQs for Hypersensitivity

Acquired C1 inhibitor deficiency

Acute generalised exanthematous pustulosis

Administration related reaction

Administration site dermatitis

Administration site eczema

Administration site hypersensitivity

Administration site rash

Administration site recall reaction

Administration site urticaria

Administration site vasculitis

Allergic bronchitis

Allergic colitis

Allergic cough

Allergic cystitis

Allergic eosinophilia

Allergic gastroenteritis

Allergic hepatitis

Allergic keratitis

Allergic oedema

Allergic otitis externa

Allergic otitis media

Allergic pharyngitis

Allergic reaction to excipient

Allergic respiratory disease

Allergic respiratory symptom

Allergic sinusitis

Allergic stomatitis

Allergic transfusion reaction

Allergy alert test positive

Allergy test positive

Allergy to immunoglobulin therapy

Allergy to surgical sutures

Allergy to vaccine

Anal eczema

Anaphylactic reaction

Anaphylactic shock

Anaphylactic transfusion reaction

Page 35 of 45

Anaphylactoid reaction

Anaphylactoid shock

Anaphylaxis treatment

Angioedema

Antiallergic therapy

Antiendomysial antibody positive

Anti-neutrophil cytoplasmic antibody positive vasculitis

Application site dermatitis

Application site eczema

Application site hypersensitivity

Application site rash

Application site recall reaction

Application site urticaria

Application site vasculitis

Arthritis allergic

Aspirin-exacerbated respiratory disease

Atopic cough

Atopy

Blepharitis allergic

Blood immunoglobulin E abnormal

Blood immunoglobulin E increased

Bromoderma

Bronchospasm

Catheter site dermatitis

Catheter site eczema

Catheter site hypersensitivity

Catheter site rash

Catheter site urticaria

Catheter site vasculitis

Chronic eosinophilic rhinosinusitis

Chronic hyperplastic eosinophilic sinusitis

Circulatory collapse

Circumoral oedema

Circumoral swelling

Conjunctival oedema

Conjunctivitis allergic

Contact stomatitis

Contrast media allergy

Contrast media reaction

Corneal oedema

Cutaneous vasculitis

Dennie-Morgan fold

Dermatitis

Dermatitis acneiform

Dermatitis allergic

Dermatitis atopic

Dermatitis bullous

Dermatitis contact

Dermatitis exfoliative

Dermatitis exfoliative generalised

Dermatitis herpetiformis

Dermatitis infected

Dermatitis psoriasiform

Device allergy

Dialysis membrane reaction

Distributive shock

Documented hypersensitivity to administered product

Drug eruption

Drug hypersensitivity

Drug provocation test

Drug reaction with eosinophilia and systemic symptoms

Eczema

Eczema infantile

Eczema nummular

Eczema vaccinatum

Eczema vesicular

Eczema weeping

Encephalitis allergic

Encephalopathy allergic

Eosinophilic granulomatosis with polyangiitis

Epidermal necrosis

**Epidermolysis** 

Epidermolysis bullosa

Epiglottic oedema

Erythema multiforme

Erythema nodosum

Exfoliative rash

Eye allergy

Eye oedema

Eye swelling

Eyelid oedema

Face oedema

Fixed eruption

Giant papillary conjunctivitis

Gingival oedema

Gingival swelling

Gleich's syndrome

Haemorrhagic urticaria

Hand dermatitis

Henoch-Schonlein purpura

Henoch-Schonlein purpura nephritis

Heparin-induced thrombocytopenia

Hereditary angioedema

Hereditary angioedema with C1 esterase inhibitor deficiency

Hypersensitivity

Hypersensitivity myocarditis

Hypersensitivity pneumonitis

Hypersensitivity vasculitis

Idiopathic urticaria

Immediate post-injection reaction

Immune thrombocytopenic purpura

Immune tolerance induction

Implant site dermatitis

Implant site hypersensitivity

Implant site rash

Implant site urticaria

Incision site dermatitis

Incision site rash

Infusion related hypersensitivity reaction

Infusion related reaction

Infusion site dermatitis

Infusion site eczema

Infusion site hypersensitivity

Infusion site rash

Infusion site recall reaction

Infusion site urticaria

Infusion site vasculitis

Injection related reaction

Injection site dermatitis

Injection site eczema

Injection site hypersensitivity

Injection site rash

Injection site recall reaction

Injection site urticaria

Injection site vasculitis

Instillation site hypersensitivity

Instillation site rash

Instillation site urticaria

Interstitial granulomatous dermatitis

Intestinal angioedema

Iodine allergy

Kaposi's varicelliform eruption

Kounis syndrome

Laryngeal oedema

Laryngitis allergic

Laryngospasm

Laryngotracheal oedema

Limbal swelling

Lip oedema

Lip swelling

Mast cell degranulation present

Medical device site dermatitis

Medical device site eczema

Medical device site hypersensitivity

Medical device site rash

Medical device site recall reaction

Medical device site urticaria

Mouth swelling

Mucocutaneous rash

Multiple allergies

Nephritis allergic

Nikolsky's sign

Nodular rash

Oculomucocutaneous syndrome

Oculorespiratory syndrome

Oedema mouth

Oral allergy syndrome

Oropharyngeal blistering

Oropharyngeal oedema

Oropharyngeal spasm

Oropharyngeal swelling

Palatal oedema

Palatal swelling

Palisaded neutrophilic granulomatous dermatitis

Palpable purpura

Pathergy reaction

Perioral dermatitis

Periorbital oedema

Periorbital swelling

Pharyngeal oedema

Pharyngeal swelling

Procedural shock

Pruritus allergic

Radioallergosorbent test positive

Rash

Rash erythematous

Rash follicular

Rash macular

Rash maculo-papular

Rash maculovesicular

Rash morbilliform

Rash neonatal

Rash papulosquamous

Rash pruritic

Rash pustular

Rash rubelliform

Rash scarlatiniform

Rash vesicular

Reaction to azo-dyes

Reaction to colouring

Reaction to excipient

Reaction to food additive

Reaction to preservatives

Red man syndrome

Rhinitis allergic

Scleral oedema

Scleritis allergic

Scrotal eczema

Scrotal oedema

Serum sickness

Serum sickness-like reaction

Shock

Shock symptom

SJS-TEN overlap

Skin necrosis

Skin reaction

Skin test positive

Solar urticaria

Solvent sensitivity

Stevens-Johnson syndrome

Stoma site hypersensitivity

Stoma site rash

Swelling face

Swelling of eyelid

Swollen tongue

Symmetrical drug-related intertriginous and flexural exanthema

Therapeutic product cross-reactivity

Tongue oedema

Toxic epidermal necrolysis

Toxic skin eruption

Tracheal oedema

Type I hypersensitivity

Type II hypersensitivity

Type III immune complex mediated reaction

Type IV hypersensitivity reaction

Urticaria

Urticaria cholinergic

Urticaria chronic

Urticaria contact

Urticaria papular

Urticaria physical

Urticaria pigmentosa

Urticaria vesiculosa

Urticarial dermatitis

Urticarial vasculitis

Vaccination site dermatitis

Vaccination site eczema

Vaccination site exfoliation

Vaccination site hypersensitivity

Vaccination site rash

Vaccination site recall reaction

Vaccination site urticaria

Vaccination site vasculitis

Vaccination site vesicles

Vaginal exfoliation

Vaginal ulceration

Vasculitic rash

Vernal keratoconjunctivitis

Vessel puncture site rash

Vessel puncture site vesicles

Vulval eczema

Vulval ulceration

Vulvovaginal rash

Vulvovaginal ulceration

Vulvovaginitis allergic

#### List of PTs under the narrow SMQs for Anaphylactic Reaction

Anaphylactic reaction

Anaphylactic shock

Anaphylactic transfusion reaction

Anaphylactoid reaction

Anaphylactoid shock

Circulatory collapse

Dialysis membrane reaction

Kounis syndrome

Procedural shock

Shock

Shock symptom

Type I hypersensitivity

#### **List of PTs for Pancreatitis**

Alcoholic pancreatitis

Autoimmune pancreatitis

Cytomegalovirus pancreatitis

Haemorrhagic necrotic pancreatitis

Hereditary pancreatitis

Immune-mediated pancreatitis

Ischaemic pancreatitis

Lupus pancreatitis

Obstructive pancreatitis

Oedematous pancreatitis

Pancreatitis

Pancreatitis acute

Pancreatitis bacterial

Pancreatitis chronic

Pancreatitis fungal

Pancreatitis haemorrhagic

Pancreatitis helminthic

Pancreatitis mumps

Pancreatitis necrotising Pancreatitis relapsing Pancreatitis viral Radiation pancreatitis Traumatic pancreatitis

#### **List of PTs for Thrombosis**

Administration site thrombosis

Adrenal thrombosis

Aortic thrombosis

Application site thrombosis

Arterial bypass thrombosis

Arterial thrombosis

Arteriovenous fistula thrombosis

Arteriovenous graft thrombosis

Atrial thrombosis

Axillary vein thrombosis

Basilar artery thrombosis

Brachiocephalic vein thrombosis

Brain stem thrombosis

Cardiac ventricular thrombosis

Carotid artery thrombosis

Catheter site thrombosis

Cavernous sinus thrombosis

Cerebellar artery thrombosis

Cerebral artery thrombosis

Cerebral thrombosis

Cerebral venous sinus thrombosis

Cerebral venous thrombosis

Coronary artery thrombosis

Coronary bypass thrombosis

Deep vein thrombosis

Deep vein thrombosis postoperative

Device related thrombosis

Foetal placental thrombosis

Graft thrombosis

Hepatic artery thrombosis

Hepatic vascular thrombosis

Hepatic vein thrombosis

Implant site thrombosis

Infective thrombosis

Infusion site thrombosis

Injection site thrombosis

Instillation site thrombosis

Intrapericardial thrombosis

Jugular vein thrombosis

Medical device site thrombosis

Mesenteric artery thrombosis

Mesenteric vein thrombosis

Ophthalmic artery thrombosis

Ophthalmic vein thrombosis

Ovarian vein thrombosis

Paraneoplastic thrombosis

Pelvic venous thrombosis

Penile vein thrombosis

Peripheral artery thrombosis

Portal vein thrombosis

Portosplenomesenteric venous thrombosis

Postoperative thrombosis

Postpartum thrombosis

Postpartum venous thrombosis

Precerebral artery thrombosis

Prosthetic cardiac valve thrombosis

Pulmonary artery thrombosis

Pulmonary embolism

Pulmonary thrombosis

Pulmonary venous thrombosis

Renal artery thrombosis

Renal vascular thrombosis

Renal vein thrombosis

Retinal artery thrombosis

Retinal vascular thrombosis

Retinal vein thrombosis

Shunt thrombosis

Spinal artery thrombosis

Splenic artery thrombosis

Splenic thrombosis

Splenic vein thrombosis

Stoma site thrombosis

Subclavian artery thrombosis

Subclavian vein thrombosis

Superior sagittal sinus thrombosis

Thrombosis

Thrombosis corpora cavernosa

Thrombosis in device

Thrombosis mesenteric vessel

Thrombosis prophylaxis

Transverse sinus thrombosis

Truncus coeliacus thrombosis

Tumour thrombosis

Umbilical cord thrombosis

Vaccination site thrombosis

Vascular access site thrombosis
Vascular graft thrombosis
Vascular pseudoaneurysm thrombosis
Vascular stent thrombosis
Vena cava thrombosis
Venous thrombosis
Venous thrombosis in pregnancy
Venous thrombosis limb
Venous thrombosis neonatal
Vertebral artery thrombosis
Vessel puncture site thrombosis
Visceral venous thrombosis